CLINICAL TRIAL: NCT02712840
Title: Pregnancy Outcomes in Good Prognosis Patients Utilizing Fresh Single Blastocyst Transfer vs. 'Freeze-All' and Delayed Frozen Single Blastocyst Transfer
Brief Title: Comparing Pregnancy Outcomes in Good Prognosis Patients Between Fresh and 'Freeze-All' Single Blastocyst Transfers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment challenge
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Ellen Greenblatt, Associate Professor; Head - Division of Reproductive Sciences; Clinical Director - Centre for Fertility and Reproductive Health, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-0167-A
Record Dates: First submitted 2015-09-09; First posted 2016-03-18 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Infertility
Keywords: Single embryo transfer; Freeze-all; Fresh; Vitrification; Clinical Pregnancy; Blastocyst
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Freeze-All Protocol (Experimental): Participants freezing all good quality embryos, with subsequent frozen embryo transfer of best quality blastocyst.
  Interventions: Procedure: Freeze-All Protocol
- Fresh Protocol (Active Comparator): Participants receiving fresh embryo transfer of best quality blastocyst and freezing of all good quality supernumerary embryos.
  Interventions: Procedure: Fresh Protocol

INTERVENTIONS:
Procedure: Freeze-All Protocol — All good morphologic quality blastocysts are vitrified on day 5 or 6. The best quality vitrified blastocyst frozen on day 5 will be warmed and transferred in a subsequent cycle.
  Arms: Freeze-All Protocol
Procedure: Fresh Protocol — Participants receive fresh embryo transfer of best morphologic quality blastocyst on day 5 and vitrification of all good quality supernumerary blastocysts.
  Arms: Fresh Protocol

SUMMARY:
The purpose of this study is to determine whether the chances of becoming pregnant are better when day the single best day 5 embryo (blastocyst) resulting from an in vitro fertilization (IVF) cycle is transferred into the uterus immediately, or after freezing the embryo and transferring it into the uterus in a subsequent cycle, separate from the ovarian stimulation used in the IVF cycle. The investigators hypothesize that in good-prognosis patients, vitrified-warmed elective single embryo transfer will result in higher implantation, clinical and on-going pregnancy and live birth rates than fresh elective single embryo transfer at the blastocyst stage.

DETAILED DESCRIPTION:
This will be a randomized controlled trial involving good prognosis infertility patients undergoing in vitro fertilization (IVF) +/- intracytoplasmic sperm injection (ICSI). Good prognosis is defined as: age <35 years, 1st IVF or IVF/ICSI cycle, normal ovarian reserve parameters (antral follicle count (AFC) >12, antimullerian hormone (AMH) > 15 pmol/L, cycle day 3 follicle stimulating hormone (FSH) < 10 IU), primarily tubal factor/male factor with ejaculated sperm or unexplained infertility, who achieve 3 or more high quality blastocysts (adequate quality for either fresh embryo transfer or cryopreservation by 5 days post-oocyte-retrieval).

All participants will be undergoing an IVF/ICSI cycle utilizing either long gonadotropin releasing hormone (GnRH) agonist or GnRH antagonist protocols. In the long GnRH agonist cycles, participants will take a combined oral contraceptive pill (OCP) for 21-42 days. The GnRH agonist buserelin acetate (0.2 mg subcutaneously daily) will be started 5 days before the last OCP is taken, for a 5-day overlap, and continued until the day of hCG trigger. In the GnRH antagonist cycles, women will either be down-regulated with an oral combined contraceptive pill (OCP) for 14-21 days, starting on cycle day 3 of the pre-stimulation cycle, or with estrogen 4 mg orally daily starting approximately 7 days post-ovulation in the pre-stimulation cycle. Participants continue the OCP or estrogen until the designated stop day as determined by the clinic schedule. In both agonist and antagonist cycles, FSH will be given to each patient in either recombinant or human menopausal gonadotropin (HMG) forms, at doses ranging from 150 IU (international units) to 300 IU daily, as per investigator judgment. FSH will start on either a natural day 3 following OCP or estrogen withdrawal, or on an 'assigned' day 3, based on scheduling requirements. The FSH dose will be maintained for 4 days, after which dose titration can occur according to results of follicular development seen on transvaginal ultrasonography and serum estradiol levels, which first occurs on cycle day 7. Continued ultrasonographic and serum level monitoring will occur every 1-2 days until time of human chorionic gonadotropin (hCG) trigger. In the GnRH antagonist cycles, a GnRH agonist will be started at a dose of 250 mcg daily when any of the following first occurs: cycle day 9, estradiol level > 2000 pmol/L, lead follicle > 14 mm in diameter, and will be continued until time of hCG trigger. Timing of hCG (5000-10,000 IU) administration will occur once at least three lead follicles have diameters > 17 mm. Oocyte retrieval will be performed 36 hours after hCG administration.

Fertilization will utilize either routine IVF or ICSI, depending upon the etiology of infertility and the quality of sperm. With ICSI, only mature oocytes will be inseminated. Embryo evaluation will occur per the clinic's standard protocols. Embryo assessment on day 5 post-fertilization will dictate final eligibility for study enrollment. Consenting participants with 3 or more cryopreservation-quality blastocysts (2BB or higher, graded according to Gardner's criteria) will then be randomized to either fresh single embryo transfer (SET) (and cryopreservation of all good quality supernumerary blastocysts) or a single frozen embryo transfer (FET) delayed to the subsequent menstrual cycle following cryopreservation of all of the good quality blastocysts. All FET cycles will be performed under a standard endometrial preparation protocol involving vaginal estradiol administration for approximately 14 days. Luteal support in either fresh or FET cycles will be with vaginal micronized progesterone, 200 mg vaginally 2-3 times daily, starting the day following fresh ET, and 6 days prior to FET, once documented endometrial thickness of 8 mm or more is achieved. The best quality blastocyst will be transferred first. Should the best blastocyst not survive warming in the FET group, the second-best blastocyst will be used. All cryopreservation will be performed by vitrification. Luteal phase progesterone will continue until either 10 weeks gestation (in an ongoing pregnancy) or until a documented negative serum hCG level drawn 14 days after the date of embryo transfer.

With a documented positive hCG serum level, the participant will undergo a transvaginal ultrasound at 7 weeks gestation to document number of gestational sacs (implantation) and clinical pregnancy rate (positive fetal heart beat). Confirmation of ongoing pregnancy (beyond 12 weeks gestation) will be obtained by review of hospital records for ultrasounds performed for nuchal translucency measurements or anatomic assessment.

Randomization at the blastocyst stage is chosen to avoid cycle cancellation if randomized earlier. All participants will be randomized by an intention to treat approach. All other components of the IVF/ICSI cycle including stimulation medications, monitoring protocols, etc. will be at the discretion of the participant's primary IVF physician; while this information will be documented it will not constitute criteria for enrollment.

Each successive enrolled participant to be randomized will choose a sequentially numbered, opaque, sealed envelope and be assigned to either the freeze-all or fresh transfer groups, based upon the envelope contents derived using computer generated block randomization, utilizing random block sizes of 4 and 6 participants, with a 1:1 allocation. The envelop contents will be provided by an independent individual not involved in study recruitment or clinical care of the participants.

ELIGIBILITY:
Inclusion Criteria:

* First IVF cycle
* Normal ovarian reserve parameters (antral follicle count > 12, follicle stimulating hormone (FSH) < 10 IU/L, AMH (if measured) > 15 pmol/L)
* Infertility cause due to tubal factor, male factor with ejaculated sperm or unexplained
* 3 or more fresh transfer or cryopreservation-quality blastocysts on day 5 post-oocyte-retrieval
* GnRH antagonist or long GnRH agonist cycles

Exclusion Criteria:

* Evidence of (or evidence for significant risk of) ovarian hyperstimulation syndrome (OHSS) on post-oocyte-retrieval day 5 (in which the standard protocol is not to perform a fresh embryo transfer, but rather to freeze all blastocysts for future frozen embryo transfers).
* Use of a gonadotropin releasing hormone (GnRH) agonist trigger for ovulation and resulting intensive luteal phase support protocol.
* Women requiring automatic freeze-all approaches (such as for pre-implantation genetic testing or cryopreservation for fertility preservation).
* Female infertility causes that may adversely affect implantation, such as severe endometriosis, fibroids, mullerian abnormalities, or prior uterine procedures resulting in a potentially compromised endometrial cavity.
* In-vitro maturation of oocytes
* Oocyte donation cycles

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2015-09; Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks of gestation
  Ongoing pregnancy is a pregnancy with a positive heart beat beyond 12 weeks of gestation.

SECONDARY OUTCOMES:
Implantation rate | 4-5 weeks after date of embryo transfer
  Implantation rate is the number of gestational sacs seen via transvaginal ultrasonography 4-5 weeks after embryo transfer, per number of embryos transferred.
Clinical pregnancy rate | 4-5 weeks after date of embryo transfer
  Clinical pregnancy is the presence of a gestational sac seen by transvaginal ultrasonography 4-5 weeks after embryo transfer.
Cumulative implantation rate | 4-5 weeks after date of blastocyst transfer
  Implantation rate for all blastocysts transferred from the same ovarian hyperstimulation IVF cycle. Includes all blastocysts transferred fresh and/or vitrified (depending upon arm of study).
Cumulative clinical pregnancy rate | 4-5 weeks after the date of blastocyst transfer
  Clinical pregnancy rate for all blastocysts transferred from the same ovarian hyperstimulation IVF cycle. Includes all blastocysts transferred fresh and/or vitrified (depending upon arm of study).
Cumulative ongoing pregnancy rate | 12 weeks of gestation for each pregnancy achieved
  Ongoing pregnancy rate for all blastocysts transferred from the same ovarian hyperstimulation IVF cycle. Includes all blastocysts transferred fresh and/or vitrified (depending upon arm of study).
Live birth rate | 10 months post-blastocyst transfer
  Number of live births achieved per blastocyst transfer
Cryopreservation thaw rate | 12 months
  Percentage of vitrified blastocysts which survive warming

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Greenblatt, MD CM, Principal Investigator — Mount Sinai Hospital, University of Toronto; Jason E Elliott, MD, MSc, Study Director — Mount Sinai Hospital, University of Toronto
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada